CLINICAL TRIAL: NCT06695260
Title: Diagnosing Dynamic Scapholunate Instability with Computer Tomography
Acronym: stressct
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Regionaal Ziekenhuis Heilig Hart Tienen (Other)
Responsible Party: Principal Investigator, Goorens Chul Ki, principal investigator, medical doctor, Regionaal Ziekenhuis Heilig Hart Tienen
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: RZ T EC 109; EC 109 (Other: RZ Tienen)
Record Dates: First submitted 2024-11-14; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Scapholunate Dissociation
Keywords: dynamic; scapholunate; instability; CT
MeSH Terms: interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Intervention Model Description: Part 1:
  To assess the normal dynamics of the scapholunate joint in patients without scapholunate instability with CT when the wrist is under loading compared to normal conditions
  Part 2:
  To assess the dynamic character of the scapholunate joint in patients with scapholunate instability with CT when the wrist is under loading compared to normal conditions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- patients with scapholunate instability (Experimental): to assess the dynamic character of the scapholunate joint in patients with scapholunate instability
  Interventions: Diagnostic Test: CT scan

INTERVENTIONS:
Diagnostic Test: CT scan — CT will be performed when the wrist is under loading compared to normal conditions. scapholunate kinematics will be examines

SUMMARY:
Scapholunate instability can result in debilitating pain, dysfunction, and secondary arthritis. If treatment is required, the instability should ideally be addressed in the dynamic stage, before non-reducible non-repairable deformation occurs. Early diagnosing of instability of the scapholunate joint can be a complex task.

In this study, the use of computer tomography (CT) scan is evaluatedto reveal the dynamic characteristics of the scapholunate instability. A CT-scan will be performed of the non-stressed wrist and a CT-scan under loading to potentially visualize increase of dorsal scaphoid translation, which is considered as primary cause of dorsoradial radioscaphoid pain in the early stage of scapholunate instability.

DETAILED DESCRIPTION:
Part 1: Assessment of the normal scapholunate stability with CT scan with and without loading in patients without symptoms of scapholunate instability

40 patients without scapholunate instability, with normal scaphoid shift test will be included. Radiographs of both wrists will be performed (anteroposterior view in pronation, clenched fist in pronation, ulnar deviation + clenched fist in supination and a sagittal view). Measurements will be the scapholunate, radiolunate, capitolunate angle and the radioscaphoid distance/angle. Then, they will undergo CT scan of both wrists without loading of the wrists (full pronation). Then, a CT scan of both wrists with loading of the wrists (supination, ulnar deviation and clenched fist) will be performed. Segmentation of the CT scans will be performed to be able to compare both CT scans. The measurements will be scapholunate distance, radioscaphoid distance, radiolunate distance, radioscaphoid rotation, radiolunate rotation and scapholunate rotation.

Exclusion criteria: <18 years, arthritis, previous wrist disorders

Part 2: Assessment of the scapholunate instability with CT scan with and without loading in patients with symptoms of scapholunate instability

40 patients with scapholunate instability, with positive scaphoid shift test will be included. Radiographs of both wrists will be performed (anteroposterior view in pronation, clenched fist in pronation, ulnar deviation + clenched fist in supination and a sagittal view). Measurements will be the scapholunate, radiolunate, capitolunate angle and the radioscaphoid distance/angle. Then, they will undergo CT scan of both wrists without loading of the wrists (full pronation). Then, a CT scan of both wrists with loading of the wrists (supination, ulnar deviation and clenched fist) will be performed. Segmentation of the CT scans will be performed to be able to compare both CT scans. The measurements will be scapholunate distance, radioscaphoid distance, radiolunate distance, radioscaphoid rotation, radiolunate rotation and scapholunate rotation. MRI scan will be performed to reveal the ligament attenuation of the scapholunate complex.

Treatment options will be proposed as usual: conservative (medication, physiotherapy) and surgery (arthroscopic capsuloligamentous repair). If arthroscopy is agreed, arthroscopic assessment of the ligamentous complex will be performed.

Correlation of the CT findings will be performed with the MRI and arthroscopic findings.

Exclusion criteria: <18 years, arthritis, previous wrist disorders

ELIGIBILITY:
Inclusion Criteria:

* >18 years

Exclusion Criteria:

* Associated fractures or other lesions

  * Neurological and severe psychological disorders
  * History of ipsilateral wrist disorders
  * Substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
dorsal radioscaphoid translation | preop assessment
  the translation of the scaphoid due to the instability is measured

SECONDARY OUTCOMES:
scapholunate distance | preop assessment
  scapholunate distance
scapholunate angle | preop assessment
  scapholunate angle in sagital view

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Scheerlinck, clinical professor, Study Chair — Universitair Ziekenhuis Brussel
Locations (1):
- Regionaal Ziekenhuis Tienen, Boutersem, Belgium

IPD SHARING:
Plan to Share IPD: No